CLINICAL TRIAL: NCT01289847
Title: A Phase IV, Multicenter, Open-Label Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Gammaplex in Primary Immunodeficiency Diseases (PID) in Children and Adolescents
Brief Title: A Study to Find Out How Safe and Effective Gammaplex® is in Young People With Primary Immunodeficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GMX04; IND 12569 (Registry Identifier: CBER)
Record Dates: First submitted 2011-01-27; First posted 2011-02-04 (Estimated); Results first posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Primary Immune Deficiency Disorders; Common Variable Immunodeficiency; X-linked Agammaglobulinemia; Hyper-IgM Syndrome; Wiskott-Aldrich Syndrome
Keywords: Primary Immune Deficiency Disorders; Common Variable Immunodeficiency; X-linked agammaglobulinemia; Hyper-IgM syndrome; Wiskott-Aldrich Syndrome; Immunoglobulins; Bacterial Infections
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Common Variable Immunodeficiency; Bruton type agammaglobulinemia; Hyper-IgM Immunodeficiency Syndrome; Wiskott-Aldrich Syndrome; Bacterial Infections | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gammaplex (Experimental)
  Interventions: Biological: Gammaplex

INTERVENTIONS:
Biological: Gammaplex — GAMMAPLEX 5g/100 mL, dose is 300-800 mg/kg/infusion every 21 or 28 days, intravenously. The total duration of treatment with GAMMAPLEX will be 12 months with a 3 month follow-up.

SUMMARY:
The main objective is to determine the efficacy of Gammaplex by measuring the number of serious acute bacterial infections during treatment with Gammaplex over a 12 month period. The secondary objectives are to assess the safety and tolerability of Gammaplex and to compare the data collected from adult subjects with PID from the GMX01 study

ELIGIBILITY:
Inclusion Criteria:

* The subject is between the ages of or is equal to 2 and 16 years of age, of either sex, belonging to any ethnic group, and above a minimum weight of 10 kg. This weight is based on the amount of blood required for testing.
* The subject has a primary immunodeficiency disease, which has as a significant component of hypogammaglobulinemia and/or antibody deficiency (e.g. common variable immunodeficiency, X-linked and autosomal forms of agammaglobulinemia, hyper-IgM syndrome, Wiskott-Aldrich Syndrome). NB Isolated deficiency of a single IgG subclass, or of specific antibodies without hypogammaglobulinemia per se, does not qualify for inclusion.
* Subjects already receiving IGIV replacement therapy require the following before their first infusion of Gammaplex:
* Documented IGIV dose(s) and treatment intervals for the last 2 consecutive routine IGIV treatments (one of which can be the screening visit result). The previous doses should also meet the following conditions before study entry: Have not changed by ± 50% of the mean dose for at least 3 months; be between 300 and 800 mg/kg/infusion; be given every 21-28 days, inclusive; be a licensed or investigational product (Phase III or IIIb).
* Documented previous IgG trough levels for the last 2 consecutive routine IGIV treatments for the last 2 consecutive routine IGIV treatments: Maintained at least 300 mg/dL above baseline serum IgG levels (defined as before initiation of any gamma globulin treatment for that subject); must be more than/equal to 600 mg/dL.
* If a subject is a female of child-bearing potential, she must have a negative result on an HCG-based pregnancy test.
* If a subject is a female who is or becomes sexually active, she must practice contraception by using a method of proven reliability for the duration of the study.
* The subject is willing to comply with all aspects of the protocol, including blood sampling, for the duration of the study.
* The subject, if old enough (generally 6 years to 16), has signed a Child Assent Form and the subject's parent or legal guardian has signed the Informed Consent Form, both approved by the IEC/IRB.

Exclusion Criteria:

* Has not been treated with IGIV (treatment naive subject)
* The subject has a history of any severe anaphylactic reaction to blood or any blood-derived product.
* The subject is known to be intolerant to any component of Gammaplex, such as sorbitol (i.e. intolerance to fructose).
* The subject has selective IgA deficiency, history of reaction to products containing IgA, or has a history of antibodies to IgA.
* Subjects who have completed the study and subjects who have withdrawn cannot participate in the study for a second time.
* The subject is currently receiving, or has received, any investigational agent, other than an immune serum globulin (ISG) preparation that is being evaluated in a Phase III or IIIb study, within the prior 3 months.
* The subject has been exposed to blood or any blood product or derivative within the last 6 months, other than a commercially available IGIV or other forms of commercially available and licensed ISG. If an unlicensed ISG product that is in Phase III or IIIb has been given, the subject cannot be infused with Gammaplex until 20 days after the last dose was given.
* The subject is pregnant or is nursing.
* The subject, at screening, has levels greater than 2.5 times the upper limit of normal as defined at the central laboratory of any of the following: (Alanine transaminase (ALT); Aspartate transaminase (AST) Lactate dehydrogenase (LDH)).
* The subject has a severe renal impairment (defined as serum creatinine greater than 2 times the upper limit of normal or BUN greater than 2.5 times the upper limit of normal for the range of the laboratory doing the analysis); the subject is on dialysis; the subject has a history of acute renal failure.
* The subject is known to abuse alcohol, opiates, psychotropic agents, or other chemicals or drugs, or has done so within the past 12 months.
* The subject has a history of DVT, or thrombotic complications of IGIV therapy.
* The subject suffers from any acute or chronic medical condition (e.g. renal disease or predisposing conditions for renal disease, or protein losing state) that, in the opinion of the investigator, may interfere with the conduct of the study.
* The subject has an acquired medical condition, such as, chronic or recurrent neutropenia (ANC < 1000 x 109/L) or AIDS known to cause secondary immune deficiency, or is post or recovering from hematopoietic stem cell transplantation.
* The subject is receiving the following medication: Systemic long-term corticosteroids (i.e. not intermittent or burst, daily, >1 mg of prednisone equivalent/kg/day).
* The subject is receiving Immunosuppressive or Immunomodulatory drugs.
* The subject has non-controlled arterial hypertension.
* The subject has anemia (hemoglobin <10 g/dL) at screening.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim J. Aldwinckle, MD, Study Director — Medical Director
Locations (10):
- United States (8):
  - Department of Medicine, University of California, Irvine, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - IMMUNOe International Reseach Centers, Centennial, Colorado
  - Family Allergy & Asthma Center, PC, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Allergy, Asthma & Immunology Clinic, P.A, Irving, Texas
  - Children's Hospital of Richmond, VA, Richmond, Virginia
- Hospital de Niňos Roberto del Río, Santiago, Chile
- Safra Children's Hospital, Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Derived] Geng B, Clark K, Evangelista M, Wolford E. Low rates of headache and migraine associated with intravenous immunoglobulin infusion using a 15-minute rate escalation protocol in 123 patients with primary immunodeficiency. Front Immunol. 2023 Feb 2;13:1075527. doi: 10.3389/fimmu.2022.1075527. eCollection 2022. PMID 36818468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First enrollment: 06 April 2011; Last Subject completed 23 April 2014; Nine recruiting sites globally: United States (US) (seven sites), Chile (one site) and Israel (one site)
Pre-assignment Details: This was a Phase IV, multicentre, open-label, non-randomised study. All enrolled subjects received study medication.
Period: Overall Study
Arm/Group | Gammaplex
Started | 25
Completed | 24
Not Completed | 1
Not completed — Patient could not comply with visits | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gammaplex
Number analyzed (Participants) | 25
Age, Customized [Number; unit: participants]
  2 to 5 year age group | 3
  6 to 11 year age group | 12
  12 to 16 year age group | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 22
  Israel | 2
  Chile | 1

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of subjects with serious, acute, bacterial infections as a measure of efficacy
Time Frame: 12 months
Population: Intent to Treat (ITT)
Measure: Number; unit: participants
Arm/Group | Gammaplex
Number analyzed (Participants) | 25
participants | 2
Statistical Analysis 1: Comparison: Gammaplex; For the primary efficacy analysis, the SABI rate for GAMMAPLEX and the upper bound of its one-sided 99% confidence interval (CI) were estimated by using the exact method for a one-sample Poisson rate; Test type: Superiority or Other; p = 0.01, one-sample Poisson rate

2. Secondary Outcome: Therapeutic Efficacy
Description: Number and proportion of subjects who maintain trough IgG levels at least as high as the average of the 2 previous trough levels before the first Gammaplex infusion
Time Frame: From week 15 onwards
Population: Seven subjects (28.0%) maintained trough IgG levels at all visits that were at least as high as the average of the two previous levels before the first infusion
Measure: Number; unit: participants
Arm/Group | Gammaplex
Number analyzed (Participants) | 25
participants | 7
Statistical Analysis 1: Comparison: Gammaplex; Test type: Superiority or Other; p = 0.01, one-sample Poisson method

3. Secondary Outcome: Therapeutic Efficacy
Description: Number of days off school
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Gammaplex
Number analyzed (Participants) | 25
days | 7.8 (12.06)

4. Secondary Outcome: Therapeutic Efficacy
Description: Number of days in hospital
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Gammaplex
Number analyzed (Participants) | 25
days | 0.3 (0.87)

5. Secondary Outcome: Therapeutic Efficacy
Description: Visits to physicians and/or emergency room
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Gammaplex
Number analyzed (Participants) | 25
visits | 4.0 (4.67)

6. Secondary Outcome: Therapeutic Efficacy
Description: Number of days on therapeutic antibiotics
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Gammaplex
Number analyzed (Participants) | 25
days | 32.0 (28.28)

ADVERSE EVENTS:
Time Frame: AEs were documented from the date Informed Consent Form or Assent was signed until 30 days after the last dose of Gammaplex was infused.
Arm/Group | Gammaplex
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gammaplex (N=25)
left lower lobe pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — A chest X-ray revealed a 4 cm retrocardiac left lung base infiltrate. Laboratory results included a WBC count of 26.4 × 109/L (ref range 4.8-10.8 × 109/L), band neutrophils 23% (ref range 50-80%) and lymphocytes 6% (ref range 20-50%). Resolved.
left lower lobe pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — The subject was hospitalised with a fever (101.8°F), tachycardia, dyspnoea, hypoxia and vomiting. No bacterial aetiology was identified by blood cultures. Resolved.
Acute Gastroenterirtis (AGE) (Gastrointestinal disorders) | 1 (1) — Three days prior to hospital admission the subject experienced watery diarrhea and vomiting. It was reported that the subject would not eat or drink and had a one-time fever of 38.1 degrees celsius. Resolved.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gammaplex (N=25)
Nasopharyngitis (Infections and infestations) | 8 (11)
Acute sinusitis (Infections and infestations) | 7 (9)
Upper respiratory tract infection (Infections and infestations) | 6 (8)
Viral upper respiratory tract infection (Infections and infestations) | 5 (7)
Pharyngitis streptococcal (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 3 (7)
Gastroenteritis viral (Infections and infestations) | 3 (4)
Pharyngitis (Infections and infestations) | 3 (4)
Bronchitis (Infections and infestations) | 2 (3)
Lobar pneumonia (Infections and infestations) | 2 (3)
Bronchitis acute (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 2 (2)
Otitis media acute (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (19)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (17)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pyrexia (General disorders) | 9 (15)
Fatigue (General disorders) | 5 (11)
Malaise (General disorders) | 5 (7)
Chest discomfort (General disorders) | 3 (6)
Infusion site erythema (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Headache (Nervous system disorders) | 13 (39)
Nausea (Gastrointestinal disorders) | 6 (8)
Vomiting (Gastrointestinal disorders) | 5 (8)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (13)
Hypotension (Vascular disorders) | 4 (12)
Diastolic hypertension (Vascular disorders) | 3 (5)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3)
Tachycardia (Cardiac disorders) | 3 (6)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the PI and Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results.

Publication of Study results will be allowed only with prior written approval from Sponsor. At the request of Sponsor, the Institution and/or Investigator shall delete any Confidential Information pertaining to Sponsor's Inventions from any proposed publications prior to submitting or presenting the materials.